CLINICAL TRIAL: NCT04467333
Title: Giessen Pulmonary Hypertension in Lung Cancer Registry
Acronym: PHLHR
Status: Recruiting | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Other Study IDs: PH in lung cancer registry
Record Dates: First submitted 2020-07-01; First posted 2020-07-13 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Hypertension Due to Lung Diseases and Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All lung cancer patients: There will not be an intervention.
  Interventions: Other: All lung cancer patients.

INTERVENTIONS:
Other: All lung cancer patients. — There will be no specific interventions. All patients will receive guidelines based therapy of lung cancer and their comorbidities.

SUMMARY:
The aim of this study is to investigate the frequency and implications of pulmonary hypertension in lung cancer patients. To do so, data will be collected from all lung cancer patients at the university hospital Giessen. All data will be analyzed for possible hints of pulmonary hypertension as a comorbidity in lung cancer patients. All information will be generated from the regular guidelines based course of treatment and there will be no interventions. This study will serve as a prospective register for all lung cancer patients treated at the university hospital Giessen.

ELIGIBILITY:
Inclusion Criteria:

* Patient with lung cancer at the University of Giessen lung Cancer Center.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Equivalent to the average of patients with lung cancer in Germany.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-06-29 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2040-01-29 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function test measured via Spirometry. | 2 years
  vital capacity, total lung capacity, forced expiratory volume in one second, functional vital capacity, diffusing capacity for carbon monoxide, arterial partial pressure of oxygen; all measured as % of predicted normal values.
sPAP values measured via Echocardiography. | 2 years
  systolic pulmonary artery pressure (sPAP) measured in millimetre of mercury (mmHg).
Body mass index. | 2 years
  weight and height will be combined to report BMI in kg/m^2.
Overall Survival and Progression Free Survival measured in days. | 2 years
  Overall Survival and Progression free survival in days will be determined by Kaplan-Meier Analysis .Measuared in (st) (time from diagnosis to death)
Measurements of the pulmonary artery diameter (PA) and ascending aorta (AA) diameter measured via computed tomography scan. PA and AA will be measured in millimeters. | 2 years
  PA and AA will be combined to report the PA/AA quotient as indicator for pulmonary hypertension in all lung cancer patients. With a cut off value of ≥ 1 defining pulmonary hypertension.
6 Minute Walk Test in meters. | 2 years
  The 6 minute walk test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance in meters covered over a time of 6 minutes is used as the outcome.
Modified Medical Research Council Scale (mMRC). | 2 years
  Scores on the mMRC reach from 0-4, with higher scores indicating greater dyspnea.
chronic obstructive pulmonary disease assessment test (CAT). | 2 years
  Scores on the CAT reach from 0-40, with higher scores indicating greater dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Bastian Eul, MD, Principal Investigator — JLU Giessen; Khodr Tello, MD, Principal Investigator — JLU Giessen
Locations (1):
- University hospital Giessen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pullamsetti SS, Kojonazarov B, Storn S, Gall H, Salazar Y, Wolf J, Weigert A, El-Nikhely N, Ghofrani HA, Krombach GA, Fink L, Gattenlohner S, Rapp UR, Schermuly RT, Grimminger F, Seeger W, Savai R. Lung cancer-associated pulmonary hypertension: Role of microenvironmental inflammation based on tumor cell-immune cell cross-talk. Sci Transl Med. 2017 Nov 15;9(416):eaai9048. doi: 10.1126/scitranslmed.aai9048. PMID 29141888
- [Derived] Rako ZA, Cekay M, Yogeswaran A, Yildiz S, Arndt PF, Kremer N, Schafer S, Janetzko P, Thal BR, Mummert CM, Franken JK, Soethe H, Werner HF, Dumitrascu R, Grimminger F, Ghofrani HA, Pullamsetti SS, Seeger W, Naeije R, Savai R, Eul B, Tello K. Echocardiographic Measure of Right Ventricular-Pulmonary Arterial Coupling Predicts Survival in Lung Cancer. Ann Am Thorac Soc. 2025 Jul;22(7):1071-1078. doi: 10.1513/AnnalsATS.202409-949OC. PMID 40042816